CLINICAL TRIAL: NCT00183755
Title: Neuroimaging Studies of Reward Processing in Depression
Brief Title: Understanding Brain Reward Responses in Individuals With Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Diego A. Pizzagalli, Associate Professor, Harvard Medical School, Mclean Hospital
Other Study IDs: R01MH068376 (NIH); R01MH068376 (NIH); DATR A3-NSS
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Depression
Keywords: Reward Processing; Anhedonia; Major Depressive Disorder; Depression
MeSH Terms: conditions — Depression; Anhedonia; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Control participants
- 2: Participants with MDD

SUMMARY:
This study will examine brain responses associated with reinforcement and reward tasks in individuals with major depressive disorder (MDD).

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a severe form of depression that can significantly interfere with an individual's thoughts, behavior, mood, and physical health. People who suffer from MDD may experience anhedonia, or the inability to gain pleasure from normally pleasurable experiences. Such individuals do not respond to motivational rewards in the same way as do individuals who are not depressed. Anhedonia has been recognized as a core symptom of depression and it is not always remedied with antidepressant medication. Abnormal brain activity and processing may be the underlying cause of depression and specifically anhedonia. A better understanding of the brain mechanisms of depression may lead to the development of new effective medications or psychological treatments.

Event-related potential (ERP), which measures electrical activity in the brain, and functional magnetic resonance imaging (fMRI), which uses scanned images to illustrate changes in brain activity, are two techniques that can identify abnormal areas of brain processing. The purpose of this study is to use ERP and fMRI to compare brain activity that is related to reward processing in individuals with MDD versus individuals without MDD.

This study will consist of 3 study visits; visits will be scheduled as close together as possible. At the first study visit, potential participants will be assessed with the SCID (Structured Clinical Interview for DSM-IV), which will identify individuals with the diagnostic criteria for MDD. A control group of non-depressed individuals will also be enrolled in the study. During the second and third study visits, participants will take part in a monetary reinforcement reward task followed by a signal detection reward task. Brain activity of all participants will be monitored during both tasks. During the second study visit, ERP will be used; during the third study visit, fMRI will be used. Demographic information will also be collected, and participants will complete several standardized questionnaires to assess mood. Some participants will be asked to return after eight weeks to complete the fMRI and EEG sessions again. Those who do complete all five sessions will be awarded a bonus.

ELIGIBILITY:
Overall Inclusion Criteria:

* Right-handed
* Agrees to use an effective form of contraception throughout the study

Inclusion Criteria for Depressed Participants:

* Meets overall inclusion criteria
* Meets DSM-IV diagnosis criteria for major depressive disorder
* Score of at least 16 on the 21-item HAM-D scale

Overall Exclusion Criteria:

* Left-handed or ambidextrous
* Claustrophobic
* Neurological or medical illness (e.g., attention deficit hyperactivity disorder, head injury, loss of consciousness, seizures)
* Pregnant

Exclusion Criteria for Depressed Participants:

* Meets any of the overall exclusion criteria
* Has been treated with electroconvulsive therapy within 6 months of study entry
* Has taken any benzodiazepine medications for at least 2 weeks prior to study entry and discontinued use of the medication for reasons other than participating in the study
* Has taken any dopaminergic medications (including methylphenidate) or neuroleptics for at least 6 months prior to study entry and discontinued use of the medication for reasons other than participating in the study
* Has taken any fluoxetine medications for at least 6 weeks prior to study entry and discontinued use of the medication for reasons other than participating in the study
* Has taken any medications that may have antidepressant properties (including some herbal supplements) within 2 weeks of study entry
* Has taken any medications that may affect blood flow (including some blood pressure medications) within 2 weeks of study entry
* Current or past history of MDD with psychotic features
* Meets DSM-IV diagnosis criteria for organic mental disorder; substance use disorder (within 1 year of study entry); lifetime substance dependence; schizophrenia; delusional disorder; bipolar disorder; post-traumatic stress disorder; eating disorder; acute bereavement; severe borderline or antisocial personality disorder; or any psychotic disorder not otherwise specified
* Current primary diagnosis of panic disorder, social phobia, generalized anxiety disorder, obsessive-compulsive disorder, or somatoform disorder

Exclusion Criteria for Control Participants

* Meets any of the overall exclusion criteria
* Diagnosed with any medical or neurological illness
* Diagnosed with any current or past psychiatric illness, as assessed by the SCID-I, including substance abuse or dependence (e.g., alcohol)
* Has taken any medications that may have antidepressant properties (including some herbal supplements) within 2 weeks of study entry
* Has taken any psychotropic medications within 2 weeks of study entry
* Has taken any medications that may affect blood flow (including some blood pressure medications) within 2 weeks of study entry

Exclusion Criteria for fMRI Studies:

* Meets any of the overall exclusion criteria
* Fails to meet safety standards for fMRI
* Current back problems
* Has strongly corrected vision, but does not wear contact lenses
* Weighs more than 250 pounds or exceeds the limit of height-to-weight ratio for a comfortable fit in the scanner
* Pregnant
* Current alcohol or substance abuse
* At risk for suicide or homicide

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Control participants, Participants with MDD
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2005-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Performance on Monetary Incentive Delay task | Given once during the second session for half an hour, and once during the third session for half an hour
  This task features balanced incentive delivery and analytic strategies designed to identify activity specific to anticipation or consumption of incentives.
Signal detection reward task | Given once during the second session for fifteen minutes, and once during the third session for fifteen minutes
  This reward task provides an objective assessment of hedonic capacity. Due to the probabilistic nature of the task, participants cannot infer which stimulus is more advantageous based on the outcome of single trials but need to integrate reinforcement history over time to optimize behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Diego A. Pizzagalli, PhD, Principal Investigator — Harvard University
Locations (3):
- United States (3):
  - The Depression Clinical and Research Program, Massachusetts General Hospital, Boston, Massachusetts
  - Affective Neuroscience Laboratory, Department of Psychology, Harvard University, Cambridge, Massachusetts
  - Athinoula A. Martinos Center for Biomedical Imaging, Massachusetts General Hospital, Charlestown, Massachusetts

REFERENCES:
- [Derived] Pizzagalli DA, Holmes AJ, Dillon DG, Goetz EL, Birk JL, Bogdan R, Dougherty DD, Iosifescu DV, Rauch SL, Fava M. Reduced caudate and nucleus accumbens response to rewards in unmedicated individuals with major depressive disorder. Am J Psychiatry. 2009 Jun;166(6):702-10. doi: 10.1176/appi.ajp.2008.08081201. Epub 2009 May 1. PMID 19411368